CLINICAL TRIAL: NCT02271698
Title: Perioperative Dexamethasone to Promote Systemic Pro-Resolution Phenotype for Prevention of Acute and Chronic Pain Post-Total Knee Arthroplasty.
Brief Title: Dexamethasone and Pain Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00055895
Record Dates: First submitted 2014-10-16; First posted 2014-10-22 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Acute Pain; Chronic Pain
Keywords: Knee arthroplasty; Dexamethasone; Acute pain; Chronic pain
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dexamethasone 6mg (Active Comparator): Patients receive 6mg iv dexamethasone at surgical incision and a repeat dose of 6mg of dexamethasone 24h after incision. Pain scores and opioid consumption will be assessed using iv opioid patient controlled analgesia totals.
  Interventions: Drug: Dexamethasone
- Dexamethasone 12mg (Active Comparator): Patients receive 12mg iv dexamethasone at surgical incision and a repeat dose of 12mg of dexamethasone 24h after incision. Pain scores and opioid consumption will be assessed using iv opioid patient controlled analgesia totals.
  Interventions: Drug: Dexamethasone
- Dexamethasone 24mg (Active Comparator): Patients receive 24mg iv dexamethasone at surgical incision and a repeat dose of 24mg of dexamethasone 24h after incision. Pain scores and opioid consumption will be assessed using iv opioid patient controlled analgesia totals.
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Patients receive a placebo injection of saline at surgical incision and a repeat placebo saline injection 24h after incision. Pain scores and opioid consumption will be assessed using iv opioid patient controlled analgesia totals.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Intravenous dexamethasone at incision and 24h after incision will be compared in 3 doses and placebo administered in a fourth group
  Other Names: Dexamethasone acetate
  Arms: Dexamethasone 12mg; Dexamethasone 24mg; Dexamethasone 6mg
Other: Placebo — Placebo injection of saline at surgical incision and a repeat placebo saline injection 24h after incision.
  Arms: Placebo

SUMMARY:
The purpose of the study is three fold. First to determine the ideal dose of dexamethasone intraoperatively that will reduce acute pain and opioid consumption. Second determine if dexamethasone at the time of surgery reduces chronic pain following total knee arthroplasty and finally determine if a pro-inflammatory environment makes patients susceptible to chronic pain after surgery and can dexamethasone alter this environment. Patients undergoing total knee arthroplasty will be randomized to four groups ( 0mg, 6mg, 12mg and 24mg dexamethasone) and assessments will be made of acute and chronic pain and quality of life measures. Blood samples will be drawn to assess Interleukin levels and for Macrophage sorting. For the primary efficacy endpoint of reduction of opioid consumption over 24 hours after surgery the dexamethasone regimen group will be compared to standard of care group using t-test. For comparisons of the secondary efficacy endpoints, t-test, Chi-square test and Fisher's Exact test will be used. Risks of this study include the risks of venipuncture and intravenous dexamethasone administration.

DETAILED DESCRIPTION:
This is a Phase IV single center, prospective, randomized, double-blind, dose response study designed to evaluate the optimum dose of dexamethasone to administer as an analgesic in total knee arthroplasty surgery. Randomization will be performed using computer software and the randomization order will be written and enclosed in envelopes in the study office. A total of 40 patients will be randomized to receive different doses of dexamethasone intravenously at induction of anesthesia with the same dose repeated 24 hours later. The dose groups are: 0mg, 6mg, 12mg, 24mg. The groups will be evenly divided into 10 subjects in each group. Patients will be cared for using established standard of care anesthetic and multi modal analgesia pathway used clinically at Duke University Medical Center. Knee arthroplasty generally occurs in patients over 65 years of age and an inclusion criteria is age 55 years or older is included in the study. Regional anesthesia is more technically challenging in morbidly obese patients. Because of an increased failure rate of regional anesthesia in morbidly obese patients an upper limit BMI of 40 is included in the study design.

Anesthetic regime. The anesthesia will be standard of care apart from the administration of the study drug.

Study Drug. After randomization the first dose of intravenous dexamethasone will be administered by the anesthesia care team immediately before surgery. The subject and study personnel will be blinded to the dose. The patient will be sedated and the study personnel will not be in the operating room. The dose will be recorded on the anesthesia record.

The second dose of dexamethasone will be prescribed by the PI. This will be prescribed electronically to be administered to the subject on the floor 24 hours after the first dose.

Surgery The surgery will proceed normally with no difference for the study.

Postoperative Pain Management Patients in all groups will receive standard of care postoperative analgesic regimen.

Blood Samples Blood will be drawn in preop holding (Time 0) for Interleukin 6, Interleukin10 and for macrophage sorting.

Blood samples will be repeated for Interleukin 6 and Interleukin10 at 10-14, 22-26 and 33-39hours after surgery.

Blood samples for macrophage sorting will be repeated at 33-39hours. The total blood collected will be 30ml on the day of surgery and 10 ml post operative day 1 for an overall total of 40cc.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo unilateral total knee arthroplasty.
* American Society of Anesthesiology (ASA) Physical Class 1-3.
* BMI <40 kg/m2

Exclusion Criteria:

* Revision surgery.
* Bilateral total knee arthroplasty.
* Unicompartmental knee arthroplasty.
* Patients with a contraindication to regional anesthesia. This includes abnormal clotting, skin infection in groin or near the back, the presence of neurological disorders or anatomical abnormalities of the vertebral column.
* Contraindications or known drug interactions with dexamethasone.
* Use of any of the following medications within the times specified before surgery:

  * Long-acting opioid medication within 3 days.
  * Any opioid medication within 24 hours.
* Body weight less than 50 kilograms (~110 pounds).
* Planned administration of another investigational product or procedure during the subject's participation in this study.
* Suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, may interfere with study assessments or compliance.
* Current or historical evidence of any clinically significant disease or condition that, in the opinion of the Investigator, may increase the risk of surgery or complicate the subject's postoperative course.
* Significant medical conditions or laboratory results that, in the opinion of the Investigator, indicate an increased vulnerability to study drugs and procedures, and expose the subject to an unreasonable risk as a result of participating in this clinical trial, such as: debilitating diseases, acute illnesses, hypotension, partial or complete conduction block, impaired cardiac function (Ejection fraction under 35%), epilepsy, myasthenia gravis), severe renal impairment (creatinine > 1.8), comorbid conditions associated with an immunocompromised status, such as blood dyscrasias, HIV/AIDS, or recent chemotherapy.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grant, MB ChB, Principal Investigator — Duke University
Locations (1):
- DUMC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 participants signed consent. 3 participants withdrew prior to randomization
Period: Overall Study
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Started | 11 | 10 | 10 | 11
Completed | 11 | 10 | 10 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 10 | 11 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.06 (8.74) | 66.56 (8.32) | 64.14 (6.43) | 69.45 (5.45) | 67.13 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 4 | 8 | 23
  Male | 4 | 6 | 6 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Pain Score
Description: Pain scores at rest and with activity using a verbal rating scales (VRS) of 0-10, where "0" represents no pain and "10" represents worst pain ever.
Time Frame: 6, 12, 18, 24, 36 hours after surgery
Population: Participants who completed pain score at specified time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 11
units on a scale
  6 hour at rest | 3.09 (1.45) | 4.80 (2.20) | 3.56 (2.74) | 5.5 (2.54)
  6 hour with movement: number analyzed (Participants) | 11 | 10 | 8 | 9
  6 hour with movement | 4.36 (2.42) | 6.50 (3.10) | 5.88 (2.47) | 7.33 (1.80)
  12 hour at rest | 2.82 (1.99) | 3.50 (1.96) | 2.78 (1.86) | 5.18 (2.99)
  12 hour with movement: number analyzed (Participants) | 8 | 9 | 7 | 10
  12 hour with movement | 5.75 (2.25) | 6.11 (1.76) | 6.00 (2.77) | 7.30 (3.23)
  18 hour at rest | 1.55 (1.86) | 2.70 (2.45) | 2.56 (2.40) | 5.09 (2.39)
  18 hour with movement: number analyzed (Participants) | 9 | 7 | 8 | 10
  18 hour with movement | 4.00 (3.16) | 5.43 (2.99) | 4.63 (2.88) | 6.90 (3.00)
  24 hour at rest | 2.91 (2.34) | 3.50 (2.27) | 3.67 (2.65) | 4.09 (2.84)
  24 hour with movement: number analyzed (Participants) | 11 | 10 | 8 | 10
  24 hour with movement | 4.82 (2.68) | 6.50 (2.07) | 6.38 (2.33) | 7.20 (2.15)
  36 hour at rest: number analyzed (Participants) | 9 | 7 | 7 | 9
  36 hour at rest | 3.00 (2.24) | 3.86 (2.54) | 4.43 (2.30) | 2.89 (1.69)
  36 hour with movement: number analyzed (Participants) | 7 | 6 | 6 | 9
  36 hour with movement | 5.29 (1.60) | 7.00 (1.79) | 6.83 (2.23) | 6.33 (1.94)
Statistical Analysis 1: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.052, t-test, 2 sided — 6 hour pain at rest
Statistical Analysis 2: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.064, t-test, 2 sided — 6 hour pain with movement
Statistical Analysis 3: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.139, t-test, 2 sided; 12 hour pain at rest
Statistical Analysis 4: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.350, t-test, 2 sided — 12 hour pain at rest
Statistical Analysis 5: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.021, t-test, 2 sided — 18 hour pain at rest
Statistical Analysis 6: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.198, t-test, 2 sided — 18 hour pain with movement
Statistical Analysis 7: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.806, t-test, 2 sided; 24 hour pain at rest
Statistical Analysis 8: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.228, t-test, 2 sided — 24 hour pain with movement
Statistical Analysis 9: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.457, t-test, 2 sided — 36 hour pain at rest
Statistical Analysis 10: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.394, t-test, 2 sided — 36 hour pain with movement

2. Primary Outcome: Change in Opioid Consumption
Description: mg of morphine equivalents
Time Frame: 6, 12, 18, 24, 36 hours after surgery
Population: Participants who completed pain score at specified time-points.
Measure: Mean (Standard Deviation); unit: mg of morphine equivalents
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Number analyzed (Participants) | 11 | 8 | 9 | 11
mg of morphine equivalents
  6 hours | 21.10 (15.94) | 22.20 (23.54) | 11.77 (11.75) | 33.50 (21.84)
  12 hours | 42.24 (50.16) | 27.24 (30.03) | 54.23 (35.80) | 32.25 (30.74)
  18 hours: number analyzed (Participants) | 11 | 8 | 7 | 9
  18 hours | 20.30 (16.77) | 16.86 (16.93) | 43.16 (55.34) | 29.75 (37.12)
  24 hours: number analyzed (Participants) | 11 | 8 | 7 | 11
  24 hours | 25.50 (15.69) | 20.91 (17.93) | 25.86 (14.80) | 23.79 (21.79)
  36 hours: number analyzed (Participants) | 10 | 7 | 7 | 9
  36 hours | 27.00 (25.22) | 24.61 (17.13) | 36.43 (26.25) | 21.29 (13.59)
Statistical Analysis 1: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.181, t-test, 2 sided — 6 hours
Statistical Analysis 2: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.364, t-test, 2 sided — 12 hours
Statistical Analysis 3: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.605, t-test, 2 sided; 18 hours
Statistical Analysis 4: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.733, t-test, 2 sided; 24 hours
Statistical Analysis 5: Comparison: Dexamethasone 6mg vs Dexamethasone 12mg vs Dexamethasone 24mg vs Placebo; Test type: Superiority or Other; p = 0.600, t-test, 2 sided — 36 hours

3. Secondary Outcome: Change in Functional Status as Measured by Western Ontario and McMaster Universities Osteoarthritis Index
Description: The Western Ontario and McMaster Universities Osteoarthritis Index measures 17 items for functional limitation (score range 0-68). Higher score = higher difficulty with the task.
Time Frame: 30 days, 3 and 6 months following surgery
Population: Participants who completed questionnaire
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 11
units on a scale
  30 Days | 25 [18.5 to 34] | 29.5 [21.25 to 38.75] | 42 [33 to 43] | 30 [23.5 to 44.5]
  3 months: number analyzed (Participants) | 11 | 10 | 9 | 10
  3 months | 17 [12 to 23.5] | 32 [24.5 to 40.25] | 19 [12 to 35] | 24 [12.25 to 33.75]
  6 months: number analyzed (Participants) | 11 | 10 | 8 | 10
  6 months | 14 [7.5 to 22.5] | 24.5 [12.75 to 29.5] | 17 [11.5 to 22] | 16 [9 to 23]

4. Secondary Outcome: Change in Chronic Pain as Measured by Brief Pain Inventory Questionnaire
Description: Brief pain inventory questionnaire will be administered generating a score (0-40). Higher scores reflect higher perceived pain.
Time Frame: Baseline at enrollment, 3 months and 6 months after surgery
Population: Participants who completed questionnaire
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 10
units on a scale
  Baseline | 5 [4 to 8] | 5 [3 to 8] | 5 [2 to 6] | 4 [1.75 to 6]
  3 months | 1 [0 to 4] | 0.5 [0 to 2] | 2 [0.75 to 3] | 2 [1 to 4]
  6 months | 0 [0 to 0] | 2.5 [0 to 3.5] | 1 [0 to 2] | 0 [0 to 1.25]

5. Secondary Outcome: Change in Functional Status as Measured by Brief Pain Inventory Questionnaire
Description: Brief pain inventory questionnaire will be administered generating a score (0-70). Higher scores reflect higher perceived pain interference.
Time Frame: Baseline at Enrollment, 3 and 6 months after surgery
Population: Participants who completed questionnaire
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Number analyzed (Participants) | 11 | 10 | 9 | 10
units on a scale
  Baseline | 5 [4 to 8] | 5 [3 to 8] | 5 [2 to 6] | 4 [1.75 to 6]
  3 Months | 0 [0 to 2] | 5 [2.25 to 8] | 0 [0 to 3] | 1.5 [0 to 3]
  6 Months | 0 [0 to 1] | 1 [0 to 4.75] | 0 [0 to 1] | 0 [0 to 2]

6. Other Pre Specified Outcome: Change in Macrophage Proliferation
Description: Macrophage totals and differentiation will be assessed within patients and between groups.
Time Frame: Samples will be taken immediately pre incision and will be repeated at 33-39hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Interleukin 6 and 10 Levels
Description: Interleukin levels and the ratio will assess pro and anti inflammatory processes in the patients
Time Frame: Sample immediately prior to incision and at 10-14, 22-26 and 33-39hours after surgery.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Randomization to 6 month follow up
Arm/Group | Dexamethasone 6mg | Dexamethasone 12mg | Dexamethasone 24mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 2/10 | 5/10 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone 6mg (N=11) | Dexamethasone 12mg (N=10) | Dexamethasone 24mg (N=10) | Placebo (N=11)
urine retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
dizziness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
wound dehisence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes